CLINICAL TRIAL: NCT07272746
Title: Effects of a Social Robot Cognitive-Game Intervention in Older Adults With Mild Cognitive Impairment and Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202504063
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Dementia; Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interactive robot game (Experimental): The experimental group will participate in a 12-week interactive robot game. The interactive robot is a screen-based robot, with the main interaction area being a facial display.
  Interventions: Other: interactive robot game
- Routine care (No Intervention): The control group will receive routine care and will not undergo any specific interventions

INTERVENTIONS:
Other: interactive robot game — The experimental group will engage in robot games for 12 weeks, twice weekly, about 20 minutes per session
  Arms: interactive robot game

SUMMARY:
This study aims to evaluate the effects of interactive robot-based games on cognitive function, neuropsychiatric symptoms, and quality of life in patients with mild cognitive impairment and dementia. The investigators plan to recruit 80 participants and randomly assign them to a control group or an experimental group; the experimental group will participate in robot games for 12 weeks, while the control group will receive routine care. Data will be collected via questionnaires to investigate whether robot games can improve cognitive function, neuropsychiatric symptoms, and quality of life in patients with mild cognitive impairment and dementia.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of interactive robot games on cognitive function, behavioral and psychological symptoms, and quality of life in patients with mild cognitive impairment and dementia. The investigators plan to recruit 80 participants and randomly assign them to a control group or an experimental group. The experimental group will engage in robot games for 12 weeks, twice weekly, about 20 minutes per session, while the control group will receive usual care. All participants will complete four questionnaire assessments to investigate whether the robot games can improve cognitive function, behavioral and psychological symptoms, and quality of life in patients with mild cognitive impairment and dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 years or older
2. Diagnosed by a physician with Mild Cognitive Impairment, mild, or moderate dementia
3. Able to communicate in Mandarin or Taiwanese
4. Willing to participate and provides informed consent signed by the participant or their family member/legal representative

Exclusion Criteria:

1. Individuals who experience fear or aversion toward interactive robots or related equipment
2. Individuals with severe hearing or visual impairments that affect participation in activities
3. Individuals unable to complete the entire intervention due to unstable physical or mental conditions
4. Individuals deemed unsuitable for this study by physician assessment

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment(MoCA) | From baseline to 12 weeks after the intervention, with follow-up assessments at 1 month and 3 months post-intervention.
  MoCA is one of the primary assessment indicators that investigators expect to see improved after interactive robot game interventions. The MoCA assessment covers multiple cognitive domains including attention and concentration, executive function, memory, language ability, visuospatial skills, abstract thinking, calculation ability, and orientation. The full score is 30 points, with higher scores indicating better cognitive function.
Neuropsychiatric Inventory Questionnaire(NPI-Q) | From baseline to 12 weeks after the intervention, with follow-up assessments at 1 month and 3 months post-intervention.
  NPI-Q is one of the primary evaluation indicators investigators expect to improve after interactive robot game intervention.
  NPI-Q includes 12 items: delusions, hallucinations, agitation, depression, anxiety, abnormal motor behavior, sleep and nighttime behavior disorders, etc. Each item is scored for severity on a scale of 1-3 points, with higher scores indicating greater severity, and for caregiver distress on a scale of 0-5 points, with higher scores indicating greater distress. The total score is calculated by multiplying the severity and distress scores, with higher scores representing more severe symptoms.

SECONDARY OUTCOMES:
Quality of Life in Alzheimer's Disease(QoL-AD) | From baseline to 12 weeks after the intervention, with follow-up assessments at 1 month and 3 months post-intervention.
  Quality of life is one of the secondary outcome measures that investigators expect to improve after an interactive robot game intervention. The QoL-AD scale is rated by the person with dementia and their caregiver on a four-point scale (poor, fair, good, very good) for each item, with total scores ranging from 13 to 52 points, where higher scores indicate better quality of life.
Geriatric Depression Scale 15(GDS-15) | From baseline to 12 weeks after the intervention, with follow-up assessments at 1 month and 3 months post-intervention.
  The Geriatric Depression Scale-15 (GDS-15) is one of the secondary evaluation indicators that investigators hope will show improvement after an interactive robot game intervention. The GDS-15 is a self-administered assessment scale containing 15 items, with a total score ranging from 0 to 15 points, where higher scores indicate a greater tendency toward depression.